CLINICAL TRIAL: NCT05951595
Title: An Open-label, Randomised, Controlled, Non-inferiority Trial to Compare the Efficacy, Safety and Tolerability of a Fixed Dose Triple Artemisinin-based Combination Therapy (TACT) Artemether-lumefantrine-amodiaquine Versus First-line Artemisinin-based Combination Therapies (ACTs) for the Treatment of Uncomplicated Plasmodium Falciparum Malaria
Brief Title: A Study to Find Out if a Combination of 3 Medicines for the Treatment of Malaria Works as Well and is as Safe and Tolerable as Combinations of 2 Medicines
Acronym: FD-TACT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAL23001
Record Dates: First submitted 2023-06-19; First posted 2023-07-19 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Uncomplicated Plasmodium Falciparum Malaria
Keywords: Artemether; Lumefantrine; Amodiaquine; Artesunate; Triple Artemisinin-based Combination Therapy (TACT)
MeSH Terms: interventions — Artemether, Lumefantrine Drug Combination; amodiaquine, artesunate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Artemether-Lumefantrine-Amodiaquine (ALAQ) (Experimental): TACT group
  Interventions: Drug: Artemether-Lumefantrine-Amodiaquine (ALAQ)
- Artemether-Lumefantrine (AL) (Active Comparator): ACT 1 group
  Interventions: Drug: Artemether-Lumefantrine (AL)
- Artesunate-Amodiaquine (ASAQ) (Active Comparator): ACT 2 group
  Interventions: Drug: Artesunate-Amodiaquine (ASAQ)

INTERVENTIONS:
Drug: Artemether-Lumefantrine-Amodiaquine (ALAQ) — A new fixed-dose combination containing artemether, lumefantrine and amodiaquine (ALAQ) will be used in the trial. Each paediatric (dispersible) tablet will contain 20 mg artemether, 120 mg lumefantrine, 40 mg amodiaquine. Two formulations of (non-dispersible/hard) tablets, containing 50 mg or 60 mg artemether, 300 or 360 mg lumefantrine and 100 or 120 mg amodiaquine, will be used for adolescents or adults. The treatments will be administered in 6 doses over 3 days at H0, H8, H24, H36, H48 and H60. The target dosing will be in line with the ranges recommended by the WHO (total dose of 5-24 mg/kg of artemether, 29-144 mg/ kg of lumefantrine, 22.5-45 mg/kg of amodiaquine).
  Arms: Artemether-Lumefantrine-Amodiaquine (ALAQ)
Drug: Artemether-Lumefantrine (AL) — A fixed-dose combination of AL will be used in the trial. Each paediatric (dispersible or non-dispersible) tablet will contain 20 mg artemether, 120 mg lumefantrine and adult (non-dispersible) tablets will contain 80 mg artemether, 480 mg lumefantrine. Treatment doses will be administered in 6 doses over 3 days at H0, H8, H24, H36, H48 and H60. The target dosing will be in line with the ranges recommended by the WHO.
  Arms: Artemether-Lumefantrine (AL)
Drug: Artesunate-Amodiaquine (ASAQ) — ASAQ will also be administered as a fixed dose combination. The tablets will contain 25 mg of artesunate and 67.5 mg of amodiaquine in the paediatric formulation and 100 mg artesunate, 270 mg amodiaquine in the adult formulation. The dosing will be administered once a day for 3 days at H0, H24 and H48 according to the schedule currently recommended by the WHO.
  Arms: Artesunate-Amodiaquine (ASAQ)

SUMMARY:
The goal of this open-label randomised, controlled, non-inferiority trial is to assess and compare the efficacy, tolerability and safety of a fixed dose TACT artemether-lumefantrine-amodiaquine (ALAQ) to the ACTs artemether-lumefantrine (AL), artesunate-amodiaquine (ASAQ) (with single low-dose primaquine in some sites) for the treatment of uncomplicated Plasmodium falciparum malaria in patient. The main question it aims to answer is whether ALAQ, a fixed dose TACT, is as efficacious, safe and tolerable in comparison with AL and ASAQ.

Participants will be enrolled, admitted and randomised to receive the study drug (ALAQ, AL or ASAQ). Patients will receive directly observed treatments and will be followed up at least once daily for the first 3 days after enrolment followed by weekly visits from D7 up to D42. Patients will be asked to report to the clinics between scheduled visits in case of any illness or other symptoms or complaints.

DETAILED DESCRIPTION:
Study participants with an uncomplicated P. falciparum monoinfection complying with all the inclusion criteria and without any of the exclusion criteria will be enrolled and randomised to three arms TACT (ALAQ), ACT1 (AL), ACT2 (ASAQ) at the sites in Africa and two arms TACT (ALAQ) and ACT (AL) at the site in Asia. Competitive recruitment with overall trial sample size 1,680 subjects (840 ALAQ, 420 AL, 420 ASAQ, i.e. a 2:1:1 ratio overall). In lower transmission settings (Annual Parasite Incidence <50 per 1000 population per year) the treatment will include a single 0.25 mg/kg gametocytocidal dose of primaquine as recommended by the World Health Organization (WHO) for patients ≥10 kg. Primaquine may be given if local treatment policy includes it.

Participants will be admitted for three days to an in-patient unit for directly observed treatment and to perform all the required study procedures from D0H0 (time of first dose intake) to D3 (H72). They will be followed up weekly starting D7 up to D42.

Microscopy to detect and quantify malaria parasitaemia will be performed daily (more frequently in participants with parasite density of >5000/µL at screening) during hospitalization and at all weekly and unscheduled visits. In participants with parasite densities >5000/µL at screening, parasite clearance rates will be assessed by repeated assessments of the parasite counts after the start of the antimalarial treatments. A capillary blood sample will be taken at each of the time-points for these parasite counts.

A physical examination and measurements of vital signs along with a symptom questionnaire will be performed and recorded through a standardized method at baseline, daily during admission and weekly during follow up through D42 and at all unscheduled visits.

Safety assessments will be performed by measuring markers of renal and hepatic toxicity, haemoglobin, platelet counts, absolute and differential white blood cell counts and electrocardiographs (ECGs). ECGs will be performed during hospitalization (H0, H4, and 4 hours after the last dose) and day 42 of follow up to assess and compare the effect of the TACT and ACTs on QT or corrected QT (QTc) intervals.

Pharmacokinetic measurements will be linked to measures of efficacy and toxicity. To reduce the burden of blood draws, especially in children, a population pharmacokinetic approach requiring sparse blood sampling will be followed in a subset of participants.

Blood samples for parasite genotyping as well as genomic and transcriptomic studies will be collected at baseline and also on the day of a recurrent infection. In selected study sites, P. falciparum parasites will be cryopreserved for in vitro antimalarial drug sensitivity testing. Where possible, ex vivo or in vitro assessments of parasite susceptibility to artemisinins and partner drugs will be assessed. The in vivo and ex vivo data on artemisinin and partner drug sensitivity will potentially be used to identify new genetic or transcriptomic markers/patterns of artemisinin or partner drug resistance.

The trial has been funded by Global Health Innovative Technology Fund.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥6 months (no upper limit unless one is required by local regulations) and bodyweight ≥5 kg
* Ability to take oral medication
* Fever defined as ≥38°C tympanic temperature or a history of fever within the last 24 hours
* Acute uncomplicated P. falciparum monoinfection
* Asexual P. falciparum parasitaemia: 1,000/µL to 250,000/µL determined on a peripheral blood film
* Written informed consent by the participant, or by the parent/guardian in case of children lower than the age of consent, and assent if required (per local regulations)
* Willingness and ability of the participants or parents/guardians to comply with the study protocol for the duration of the study

Exclusion Criteria:

* Signs of severe malaria (adapted from WHO criteria)
* Patients not fulfilling criteria for severe malaria but with other indication(s) for parenteral antimalarial treatment at the discretion of the treating physician
* Haemoglobin <7 g/dL at screening
* Participants who have received artemisinin or a derivative within the previous 7 days OR lumefantrine or amodiaquine within the previous 14 days
* In applicable countries: use of seasonal malaria chemoprophylaxis (SMC) within the last 30 days
* Acute illness other than malaria requiring systemic treatment
* Severe acute malnutrition
* Known HIV, tuberculosis, severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) or other severe infection
* For women of child-bearing age: pregnant, trying to get pregnant or lactating
* History of allergy or known contraindication to any of the study drugs, including neuropsychiatric disorders and epilepsy
* Previous splenectomy
* Participation in the previous 3 months and/or ongoing follow-up for an interventional study (including FD-TACT)

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1680 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
28-day efficacy | 28 days
  28-day efficacy defined as the proportion of patients with Polymerase Chain Reaction (PCR)-corrected adequate clinical and parasitological response (ACPR) at Day 28, i.e., absence up to Day 28 of P. falciparum parasitaemia (detected by microscopy) with parasites genetically identical to those detected at baseline (as determined by PCR product length polymorphisms)

SECONDARY OUTCOMES:
28-day PCR uncorrected efficacy | 28 days
  28-day PCR uncorrected efficacy defined as the proportion of patients with absence up to Day 28 of P. falciparum parasitaemia
42-day efficacy | 42 days
  42-day efficacy defined as the proportion of patients with PCR-corrected adequate clinical and parasitological response (ACPR) at Day 42, i.e., absence up to Day 42 of P. falciparum parasitaemia (detected by microscopy) with parasites genetically identical to those detected at baseline (as determined by PCR product length polymorphisms)
42-day PCR-uncorrected efficacy | 42 days
  42-day PCR-uncorrected efficacy defined as the proportion of patients with absence up to Day 42 of P. falciparum parasitaemia
Parasite clearance half-life | 3 days
  Assessed by microscopy as primary parameter to determine parasite clearance half-life
Proportion of participants with microscopically detectable P. falciparum parasitaemia at Day 3 | 3 days
Fever clearance time | 42 days
  Fever clearance time (i.e., the time taken for the tympanic temperature to fall below 37.5°C in participants who were febrile at inclusion)
Proportion of participants with gametocytaemia | 42 days
  Proportion of participants with gametocytaemia during and after treatment stratified by presence of gametocytes at enrolment
Incidence of adverse events (AEs) | 42 days
  Incidence of AEs within the first 42 days including markers of hepatic, renal or bone marrow toxicity
Incidence of serious adverse events (SAEs) | 42 days
  Incidence of SAEs within the first 42 days including markers of hepatic, renal or bone marrow toxicity
Number of cardiotoxicity events | 42 days
  Cardiotoxicity in particular QT or QTc-interval above 500 ms at timepoint H4, H52 or H64, D42
Proportion of participants requiring retreatment due to vomiting | 1 hour after administration of each dose of the treatment
  Proportion of participants requiring retreatment due to vomiting within 1 hour after administration of the study drugs
Proportion of participants who report completing a full course of observed TACT | 3 days
  Proportion of participants who report completing a full course of observed TACT without withdrawal of consent or exclusion from study because of drug related serious adverse event
Proportion of participants who report completing a full course of observed ACT | 2 or 3 days depending on the treatment
  Proportion of participants who report completing a full course of observed ACT without withdrawal of consent or exclusion from study because of drug related serious adverse event
Peak plasma concentration | 42 days
  Peak plasma concentration (Cmax) of artemisinin-derivatives and partner drugs in ACT and TACT treated participants in correlation with pharmacodynamics measures of drug efficacy
Area under curve | 42 days
  Area under the plasma concentration versus time curve (AUC) of artemisinin-derivatives and partner drugs in ACT and TACT treated participants in correlation with pharmacodynamic measures of drug efficacy
Pharmacokinetic interactions - peak plasma concentration | 42 days
  Comparison of peak plasma concentration (Cmax) of artemisinin-derivatives and partner drugs in ACT and TACT treated participants in correlation with pharmacodynamics measures of drug efficacy
Pharmacokinetic interactions - area under curve | 42 days
  Comparison of area under the plasma concentration versus time curve (AUC) of artemisinin-derivatives and partner drugs in ACT and TACT treated participants in correlation with pharmacodynamic measures of drug efficacy
Plasma levels of partner drugs | 7 days
  Plasma levels of partner drugs in correlation with treatment efficacy and treatment arm on Day 7

OTHER OUTCOMES:
Comparison of 28-day PCR-corrected efficacy of ALAQ vs AL | 28 days
  Comparison of 28-day PCR-corrected ACPR (as defined in outcome measure 1) of ALAQ vs AL in infections with parasites carrying known and/or candidate markers of antimalarial drug resistance (mutations in pfkelch13, pfcrt, pfmdr1 and/or other markers, including those identified over the course of the study)
Comparison of 28-day PCR-uncorrected efficacy of ALAQ vs AL | 28 days
  Comparison of 28-day PCR-uncorrected efficacy (as defined in outcome measure 2) of ALAQ vs AL in infections with parasites carrying known and/or candidate markers of antimalarial drug resistance (mutations in pfkelch13, pfcrt, pfmdr1 and/or other markers, including those identified over the course of the study)
Comparison of 42-day PCR-corrected efficacy of ALAQ vs AL | 42 days
  Comparison of 42-day PCR-corrected ACPR (as defined in outcome measure 3) of ALAQ vs AL in infections with parasites carrying known and/or candidate markers of antimalarial drug resistance (mutations in pfkelch13, pfcrt, pfmdr1 and/or other markers, including those identified over the course of the study)
Comparison of 42-day PCR-uncorrected efficacy of ALAQ vs AL | 42 days
  Comparison of 42-day PCR-uncorrected efficacy (as defined in outcome measure 4) of ALAQ vs AL in infections with parasites carrying known and/or candidate markers of antimalarial drug resistance (mutations in pfkelch13, pfcrt, pfmdr1 and/or other markers, including those identified over the course of the study)
Comparison of 28-day PCR-corrected efficacy of ALAQ vs ASAQ | 28 days
  Comparison of 28-day PCR-corrected ACPR (as defined in outcome measure 1) of ALAQ vs ASAQ in infections with parasites carrying known and/or candidate markers of antimalarial drug resistance (mutations in pfkelch13, pfcrt, pfmdr1 and/or other markers, including those identified over the course of the study)
Comparison of 28-day PCR-uncorrected efficacy of ALAQ vs ASAQ | 28 days
  Comparison of 28-day PCR-uncorrected efficacy (as defined in outcome measure 2) of ALAQ vs ASAQ in infections with parasites carrying known and/or candidate markers of antimalarial drug resistance (mutations in pfkelch13, pfcrt, pfmdr1 and/or other markers, including those identified over the course of the study)
Comparison of 42-day PCR-corrected efficacy of ALAQ vs ASAQ | 42 days
  Comparison of 42-day PCR-corrected ACPR (as defined in outcome measure 3) of ALAQ vs ASAQ in infections with parasites carrying known and/or candidate markers of antimalarial drug resistance (mutations in pfkelch13, pfcrt, pfmdr1 and/or other markers, including those identified over the course of the study)
Comparison of 42-day PCR-uncorrected efficacy of ALAQ vs ASAQ | 42 days
  Comparison of 42-day PCR-uncorrected efficacy (as defined in outcome measure 4) of ALAQ vs ASAQ in infections with parasites carrying known and/or candidate markers of antimalarial drug resistance (mutations in pfkelch13, pfcrt, pfmdr1 and/or other markers, including those identified over the course of the study)
Proportions of recurrent infections with mutations | 42 days
  Proportions of recurrent infections with parasites carrying mutations known to be associated with recrudescence
Proportions of specimens collected at baseline with parasites carrying mutations | Baseline
  Proportions of specimens collected at baseline with parasites carrying mutations of known functional or operational significance (pfkelch13, pfcrt, pfmdr1, pfdhfr, pfdhps, pfplasmepsin2, and/or other parasite genetic markers associated with resistance or identified over the course of the study)
Change in haemoglobin concentration stratified for Glucose-6-Phosphate Dehydrogenase (G6PD) status/genotype | 28 days
  Change in haemoglobin concentration at day 3, 7, 28, stratified for G6PD status/genotype in participants receiving single low dose primaquine (SLD-PQ) vs those not receiving it
Comparison of transcriptomic patterns of drug sensitive and resistant parasites | 24 hours
  Comparison of levels of RNA transcription before treatment and 6, 12 and 24 hours after start of treatment between parasites with or without known or putative markers of drug resistance
Levels of RNA transcription coding for male or female specific gametocytes | 14 days
  Levels of RNA transcription coding for male or female specific gametocytes at admission up to day 14, stratified by the presence of gametocytes at enrolment
In vitro susceptibility of P. falciparum to artemisinins and partner drugs | 42 days
  In vitro susceptibility, measured as % survival after drug exposure or as half-maximal inhibitory concentration (IC50), of P. falciparum to artemisinins and partner drugs according to study sites and genotype
Ex vivo susceptibility of P. falciparum to artemisinins and partner drugs | 42 days
  Ex vivo susceptibility, measured as % survival after drug exposure or as IC50, of P. falciparum to artemisinins and partner drugs according to study sites and genotype

CONTACTS AND LOCATIONS:
Overall Officials: Mehul Dhorda, Ph.D, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit, Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand; Arjen Dondorp, Prof., Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit, Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand
Locations (1):
- Ruhuha Health Centre, Ruhuha, Eastern Province, Rwanda

IPD SHARING:
Plan to Share IPD: Yes
With participant's consent, participant's data and results from blood analyses stored in the database may be shared according to the terms defined in the Mahidol Oxford Tropical Medicine Research Unit (MORU) data sharing policy with other researchers to use in the future. All personal information will be anonymised so that no individual can be identified from their treatment records or through interviews.
Time Frame: After completion of the trial activities and reporting
Access Criteria: MORU data sharing policy
URL: https://www.tropmedres.ac/units/moru-bangkok/bioethics-engagement/data-sharing/moru-tropical-network-policy-on-sharing-data-and-other-outputs